CLINICAL TRIAL: NCT00331422
Title: A Phase II Study of Carboplatin and Paclitaxel as Neoadjuvant Chemotherapy Followed by Interval Cytoreduction in Women With Advanced Staged Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma for High-Risk Surgical Candidates or Patients Unlikely to be Optimally Surgically Cytoreduced
Brief Title: Carboplatin, Paclitaxel, and Surgery in Treating Patients With Advanced Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of available funding.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS070; UMN-0409M64006 (Other: Institutional Review Board, University of Minnesota); UMN- WCC-40 (Other: Women's Cancer Center, University of Minnesota)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer; fallopian tube cancer; Brenner tumor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin; Paclitaxel; Cytoreduction Surgical Procedures; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Who Received Treatment (Experimental): All patients receiving treatment with Paclitaxel and Carboplatin followed by surgery to remove cancerous tissue.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Procedure: cytoreductive surgery

INTERVENTIONS:
Drug: carboplatin — Carboplatin dose (milligrams (mg)) - Target Area Under the Curve (AUC) 6 x (Glomerular Filtration Rate+25) - Calvert Formula, given intravenously (IV) for 30 minutes.
  Other Names: Paraplatin
Drug: paclitaxel — Paclitaxel dose = 175 milligrams per meter squared (mg/m2) over 3 hours.
  Other Names: Taxol
Procedure: cytoreductive surgery — Surgery - tumor specimen collected for extreme drug resistant assay (EDR) and A1 assays for analysis
  Other Names: surgery; debulking

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or stopping them from dividing. Giving chemotherapy drugs before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with carboplatin before surgery works in treating patients with advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether at least 50% of patients with advanced ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer are able to achieve optimal cytoreduction (to < 1 centimeter of remaining disease) after neoadjuvant chemotherapy comprising paclitaxel and carboplatin.

Secondary

* Determine the frequency and severity of toxicity associated with this regimen in patients who are high-risk surgical candidates or in patients unlikely to achieve optimal surgical cytoreduction.
* Determine if extreme drug resistance assay profiles change after neoadjuvant chemotherapy.
* Determine how thrombospondin-1 (TSP-1), tumor protein 53 (p53), and tumor vessel density change after administration of neoadjuvant chemotherapy.
* Assess the quality of life of patients receiving neoadjuvant chemotherapy.
* Obtain estimates of tumor response after administration of neoadjuvant chemotherapy.
* Determine whether serum cancer antigen 125 (CA-125) at the time of cytoreduction is associated with the ability to optimally reduce the patients.

OUTLINE: This is an open-label study.

Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Within 4-6 weeks after the fourth course of chemotherapy, patients undergo interval cytoreductive surgery.

Patients who are unable to undergo surgery receive 2 additional courses of chemotherapy and are re-evaluated for surgery after the sixth course of chemotherapy.

Within 4 weeks after surgery, patients receive 2 additional courses of chemotherapy.

Quality of life is assessed periodically.

Tumor samples are obtained via laparoscopic or percutaneous biopsy prior to beginning chemotherapy and during interval cytoreduction. Tissue is examined by immunohistochemistry staining for p53, TSP-1, microvessel density (CD31), angiogenesis, membrane protein BCL-2, and multidrug resistant gene 1 (MDR-1). Gene array analysis and extreme drug resistant assays are also performed.

After completion of study treatment, patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of epithelial ovarian, primary peritoneal, or fallopian tube carcinoma for which no previous treatment has been given.

Patients with the following histological epithelial cell types are eligible:

* Serous adenocarcinoma
* Mucinous adenocarcinoma
* Clear cell adenocarcinoma
* Transitional cell
* Adenocarcinoma not otherwise specified
* Endometrioid adenocarcinoma
* Undifferentiated carcinoma
* Mixed epithelial carcinoma
* Malignant Brenner's tumor

  * Measurable or non-measurable disease as defined by Solid Tumor Response Criteria (RECIST) within 4 weeks of study entry
  * High-risk surgical candidate
  * Gynecologic Oncology Group (GOG) performance status 0-3
  * Absolute neutrophil count ≥ 1,500/mm^3
  * Platelet count ≥ 100,000/mm^3
  * Creatinine ≤ 1.5 mg/dL
  * Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
  * Bilirubin ≤ 1.5 times ULN
  * Serum glutamic oxaloacetic transaminase (SGOT) ≤ 3 times ULN
  * Life expectancy ≥ 12 weeks

Exclusion Criteria:

* Pregnant or nursing
* Positive pregnancy test -(Fertile patients must use effective nonhormonal contraception during and for 3 months after completion of study treatment.)
* History of another neoplasm except for non-metastatic, non-melanoma skin cancers, carcinoma in situ of the cervix, or cancer cured by surgery > 5 years prior to registration.
* Septicemia, severe infection, acute hepatitis, or severe gastrointestinal bleeding, defined as requiring blood transfusion or hospitalization at registration
* Unstable angina will not be eligible. Patients with evidence of abnormal cardiac conduction (e.g. bundle branch block, heart block) are eligible if their disease has been stable for the past six months.
* History of severe hypersensitivity or allergic reaction to study drugs, drugs formulated in Cremophor EL^®, other platinol compounds, or mannitol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Geller, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Who Received Treatment: Includes all patients enrolled and treated with at least one dose of chemotherapy (carboplatin - dose calculated per Calvert formula - given intravenously for 30 minutes and/or paclitaxel 175 milligrams per meter squared over 3 hours).
Period: Overall Study
Arm/Group | Patients Who Received Treatment
Started | 7 (Patients who met study criteria and received at least one dose of study drug.)
Completed | 2 (Completed all 6 courses of chemotherapy and had surgery to remove all tumor lesions.)
Not Completed | 5
Not completed — Did not receive entire study regimen | 5

BASELINE CHARACTERISTICS:
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: Years] | 67 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Underwent Optimal Cytoreduction After Chemotherapy
Description: These patients had their tumor(s) removed by surgery after receiving 4 cycles of chemotherapy to determine their response.
Time Frame: Week 18 (After 4 cycles of chemotherapy)
Population: Includes those patients that received 4 cycles of therapy before removal of cancerous tissue. Evaluation of overall response is not possible due to low number of patients and therefore could not obtain statistical significance.
Measure: Number; unit: Participants
Groups:
- Evaluable Patients (Received 4 Cycles of Therapy and Surgery): Includes patients treated with 4 cycles of study chemotherapy regimen and surgery.
Arm/Group | Evaluable Patients (Received 4 Cycles of Therapy and Surgery)
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Patients' Overall Tumor Response as Measured by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Best response recorded from start of treatment until after 4th cycle of treatment. Defined by the sum of Complete Responses (CR), Partial Responses (PR), and Stable Disease (SD) in patients neoadjuvant chemotherapy. CR=disappearance of all lesions, PR=>or=30% decrease in sumof all target lesins, Progressive Disease (PD) =>or =20% increase in sum of all target or any new lesions, SD=not CR, PR or PD.
Time Frame: Week 16 (4 weeks after 4th course)
Measure: Number; unit: Participants
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 7
Participants
  Partial Response | 2
  Progressive Disease | 3
  Stable Disease | 2

3. Secondary Outcome: Clinical Response Based on Serum Cancer Antigen 125 (CA-125) Concentration
Description: Ca-125 serum results compared from baseline to after patient's last treatment. This is a tumor biomarker. A decrease in results indicates a clinical response.
Time Frame: From Baseline to up to 12 weeks (4 courses of therapy)
Measure: Number; unit: Participants
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 7
Participants
  Increased Concentration | 1
  Decreased Concentration | 6

4. Secondary Outcome: Change in Drug Resistance After Neoadjuvant Chemotherapy
Description: As measured by extreme drug resistance assay - Unable to report due to tissue samples being incomplete or unsatisfactory to do laboratory testing.
Time Frame: Day 1 to Time to Surgery (Approximately Week 18)
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Thrombospondin-1 (TSP-1), p53, and Tumor Vessel Density
Description: Unable to report due to incomplete (nonviable) or unsatisfactory tissue samples.
Time Frame: Week 18 (At surgery)
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life Score of Patients Receiving Neoadjuvant Chemotherapy
Description: Functional Assessment of Cancer Therapy-Ovarian (FACT-O) Questionnaire was used to assess the impact of treatment- and disease-related factors on the quality of life of patients with ovarian cancers undergoing chemotherapy. It is a 5 point scale (from worse to best: 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much responses). Physical well-being, social/family well-being, functional well-being, emotional well-being and additional concerns questions are asked.
  Unable to evaluate; patients did not consistently complete the questionnaires.
Time Frame: Day 1, Week 12 (after 4th course) , Week 16 (4 weeks after last treatment)
Arm/Group | Patients Who Received Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 of treatment through 30 days post treatment or death, whichever came first.
Description: All events are reported; related and unrelated to study treatment.
Arm/Group | Patients Who Received Treatment
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received Treatment (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 3 (3)
Confusion (Nervous system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fistula, gastrointestinal (Gastrointestinal disorders) | 1 (1)
Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Infection (Infections and infestations) | 2 (4)
Infection, bladder (Renal and urinary disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Other, Failure to Thrive (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 2 (2)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Wound complication (Skin and subcutaneous tissue disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Who Received Treatment (N=7)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Double Vision (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infection (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Oxygen, decreased (pulmonary-atelectasis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral Edema (limb) (Blood and lymphatic system disorders) | 1 (1)
Sleep Apnea (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Tinnitus (ringing in ears) (Ear and labyrinth disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1 of the 2 evaluable patients was switched from Paclitaxel to Taxotere during the course of her treatment due to toxicity (adverse effects), but since it remains a platinum-based chemotherapy she is included in the evaluable group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes